CLINICAL TRIAL: NCT06156059
Title: Oral Bedtime Melatonin in Critically Ill Patients
Acronym: Mel-ICU
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Miguel Sanchez Garcia, Director Critical Care Department, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Mel-ICU
Record Dates: First submitted 2023-11-26; First posted 2023-12-05 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Septic Shock; Stroke Hemorrhagic; Strokes Thrombotic; Cardiac Arrest
MeSH Terms: conditions — Shock, Septic; Hemorrhagic Stroke; Thrombotic Stroke; Heart Arrest | interventions — Melatonin; Capsules

STUDY DESIGN:
Intervention Model Description: double blind randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Indistinguishable oral suspension or capsule
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Septic Shock Standard of Care (SOC) (Placebo Comparator): Placebo suspension and capsules
  Interventions: Drug: Placebo suspension or capsule
- Septic shock Oral Bedtime Melatonin (OBM) (Active Comparator): 100 mg suspension or in capsules OBM
  Interventions: Drug: Oral Bedtime Melatonin
- Resuscitated Cardiorespiratory Arrest SOC (Placebo Comparator): Placebo suspension and capsules
  Interventions: Drug: Placebo suspension or capsule
- Resuscitated Cardiorespiratory Arrest OBM (Active Comparator): 100 mg suspension or in capsules OBM
  Interventions: Drug: Oral Bedtime Melatonin
- Ischemic Stroke (SOC) (Placebo Comparator): Placebo suspension and capsules
  Interventions: Drug: Placebo suspension or capsule
- Ischemic stroke (OBM) (Active Comparator): 100 mg suspension or in capsules OBM
  Interventions: Drug: Oral Bedtime Melatonin
- Hemorraghic stroke (SOC) (Placebo Comparator): Placebo suspension and capsules
  Interventions: Drug: Placebo suspension or capsule
- Hemorrhagic stroke (OBM) (Active Comparator): 100 mg suspension or in capsules OBM
  Interventions: Drug: Oral Bedtime Melatonin

INTERVENTIONS:
Drug: Oral Bedtime Melatonin — 100 mg oral suspension or capsule given at bedtime
  Other Names: Oral melatonin
  Arms: Hemorrhagic stroke (OBM); Ischemic stroke (OBM); Resuscitated Cardiorespiratory Arrest OBM; Septic shock Oral Bedtime Melatonin (OBM)
Drug: Placebo suspension or capsule — Indistinguishable suspension or capsule
  Other Names: Placebo
  Arms: Hemorraghic stroke (SOC); Ischemic Stroke (SOC); Resuscitated Cardiorespiratory Arrest SOC; Septic Shock Standard of Care (SOC)

SUMMARY:
Oxidative stress is one of the main mechanisms causing harm in severe infection with septic shock, ischemia-reperfusion injury in resuscitated cardiac arrest and ischemic and hemorrhagic stroke.

Melatonin is a potent scavenger of the mediators of oxidative stress, oxygen and nitrogen-reactive species, which directly injure cell structures like walls and DNA and thus cause organ dysfunction.

In a previous study we have observed that high-dose oral bedtime melatonin (OBM) is associated with improved organ function in severe Covid-19 patients

DETAILED DESCRIPTION:
This is a double-blind randomized, adaptive trial in the 4 indications mentioned above giving 100 mg of OBM or placebo.

Interim analyses with pre-specified stopping rules will be performed in each sub-study for specific outcome variables collected at scheduled timelines.

Comparative organ dysfunction score (Sequential Organ Failure Evaluation-SOFA) will be done at baseline, 7, 14, and 30 days and mortality evaluated at 30 and 90 days.

For the 3 study groups enrolling stroke and resuscitated cardiac arrest patients, the modified Rankin score and the CVC (Glasgow) at 30 and 90 days will be compared.

ELIGIBILITY:
Inclusion Criteria:

* ICU stay >5 days

Exclusion Criteria:

* ominous prognosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Mortality at 90 days | Inclusion to 90 days
  All-cause mortality